CLINICAL TRIAL: NCT06600633
Title: Study of the Efficacy of Dietary Supplementation in Targeting Sleep Quality (NutriSom Study A)
Brief Title: Efficacy of Dietary Supplementation With Melatonin in Targeting Sleep Quality
Acronym: NutriSom-01A
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Nutrition, Slovenia (Nutris) (Other)
Collaborators: Faculty of Pharmacy, University of Ljubljana, Slovenia (Unknown); Faculty of health sciences, Celje, Slovenia (Unknown); CMS - Center za motnje spanja, Ljubljana, Slovenia (Unknown); Valens Int. d.o.o., Slovenija (Industry)
Responsible Party: Principal Investigator, Igor Pravst, Prof. Dr. Igor Pravst, Institute of Nutrition, Slovenia (Nutris)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KEP-4-6/2024-A; L7-50044 (Other Grant/Funding Number: Slovenian Research and Innovation Agency)
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Sleep Onset Latency; Sleep Quality
Keywords: melatonin; supplementation; sleep; sleep onset latency; actigraphy; sleep quality; sleep efficiency
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Three-period crossover study will include 30 subjects who will test three formulations with diferent melatonin dosages (placebo product without melatonin, and two products with different melatonin levels). Subjects will have 2 week intervention with each of the tested formulations with 2 week wash-out.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo product (PP) (Placebo Comparator): Active ingredient: none Instructions for use: Supplement should be consumed once per day during the intervention period, about one hour to bedtime.
  Interventions: Dietary Supplement: 14 days of intervention with Placebo Product (PP)
- Active control (AC) (Active Comparator): Active ingredient: 1 mg of melatonin per dosage Instructions for use: Supplement should be consumed once per day during the intervention period, about one hour to bedtime.
  Interventions: Dietary Supplement: 14 days of intervention with Active Control (AC)
- Test product (TP) (Experimental): Active ingredient: 0.3 mg of melatonin per dossage Instructions for use: Supplement should be consumed once per day during the intervention period, about one hour to bedtime.
  Interventions: Dietary Supplement: 14 days of intervention with Test Product (TP)

INTERVENTIONS:
Dietary Supplement: 14 days of intervention with Placebo Product (PP) — 1 spray (0 mg melatonin)
  Arms: Placebo product (PP)
Dietary Supplement: 14 days of intervention with Active Control (AC) — 1 spray (1 mg melatonin)
  Arms: Active control (AC)
Dietary Supplement: 14 days of intervention with Test Product (TP) — 1 spray (0.3 mg melatonin)
  Arms: Test product (TP)

SUMMARY:
single-center, randomized, cross over, double-blind, placebo controlled intervention study

DETAILED DESCRIPTION:
The single-center, randomized, cross over, double-blind, placebo controlled intervention study will include 30 subjects who will test the efficacy of three formulations with different dosages of melatonin on sleep quality parameters.

ELIGIBILITY:
Inclusion criteria:

* subject Informed consent form (ICF) is signed
* aged 24-65 years at the time of the signature of ICF
* suboptimal sleep quality according to Pittsburgh Sleep Quality Index (PSQI-SI): PSQI higher than 5
* no clinically significant (subthreshold) insomnia according to Pittsburgh Sleep Quality Index (PSQI-SI) (Kmetec et al., 2022): PSQI up to 9
* a body mass index (BMI) up to 32 kg/m2
* stable medications for non excluded concurrent medical conditions for six weeks prior to the screening visit
* ability to ingest oral food supplement (study product)
* willing to follow all study procedures, including attending all site visits and use of actigraphy

Exclusion criteria:

* diagnosed or subject to therapy due to sleep disorders
* acute infectious disease
* any kind of chronic pharmacological therapy with antihypertensives or antidepressants
* any kind of other pharmacological therapy that could interact with active ingredients used in the study
* pregnancy or planned pregnancy, lactation, menopause (with clinically relevant symptoms/therapy)
* use of beta-blockers
* chronic use of use of prostaglandin synthesis inhibitors (nonsteroidal anti-inflammatory drugs), such as acetylsalicylic acid and ibuprofen
* supplementation with melatonin or other food supplements intendent for sleep quality during last 2 weeks
* unwillingness to maintain caffeine abstinence after 4:00 PM during the study
* not having a mobile upper extremity for attaching an actigraph
* known alcohol and/or drug abuse
* unwillingness to comply with the maximum limit of 2 alcoholic drinks per day, and only up to 1 alcoholic drink after 6:00 PM during the study
* known lactose/gluten intolerances/food allergies
* known gastrointestinal disease
* less than 5 years after treatment for gastrointestinal cancer (stomach, duodenum or colon)
* have stomach or bowel resection
* night work (including as part of shift work)
* mental incapacity that precludes adequate understanding or cooperation
* participation in another investigational study

Ages: 24 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2025-09-17 (Estimated); Study Completion 2025-09-17 (Estimated)

PRIMARY OUTCOMES:
Change in sleep onset latency (SOL) compared to placebo | last 7 days of intervention
  Change in sleep onset latency (SOL) compared to placebo assessed by actigraphy.

SECONDARY OUTCOMES:
Changed sleep quality compared to placebo | 14 days
  Changed sleep quality compared to placebo - assessed by adapted Pittsburgh Sleep Quality Index (PSQI)
Changed sleep efficiency (SE) compared to placebo | last 7 days of intervention
  Changed sleep efficiency (SE) compared to placebo - assessed by actigraphy

CONTACTS AND LOCATIONS:
Overall Officials: Igor Pravst, Study Chair — Nutrition Institute, Ljubljana; Barbara Gnidovec Stražišar, Principal Investigator — Faculty of Health Sciences in Celje, CMS - Center za motnje spanja
Locations (1):
- CMS - Center za motnje spanja, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NutriSom project webpage: Efficacy and safety of dietary supplementation in targeting sleep quality (L7-50044) — https://nutris.org/en/projects/nutrisom